CLINICAL TRIAL: NCT05775471
Title: Neoadjuvant Combination Pembrolizumab / Enfortumab Vedotin With Adjuvant Pembrolizumab Prior to and After Radical Nephroureterectomy for High-Risk Upper Tract Urothelial Carcinoma
Brief Title: Pembrolizumab and Enfortumab Vedotin With Pembrolizumab Prior to and After Radical Nephroureterectomy for High-Risk Upper Tract Urothelial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-001932; NCI-2023-00999 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Renal Pelvis and Ureter Urothelial Carcinoma
MeSH Terms: interventions — Biopsy; Specimen Handling; enfortumab vedotin; Nephroureterectomy; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, enfortumab vedotin) (Experimental): Patients receive pembrolizumab IV and enfortumab vedotin IV on study. Patients undergo radical nephroureterectomy and receive pembrolizumab IV on study Patients also undergo MRU imaging and undergo blood, urine and tissue sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Enfortumab Vedotin; Procedure: MR Urography; Procedure: Nephroureterectomy; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood and urine collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Enfortumab Vedotin — Given IV
  Other Names: AGS 22ME; AGS-22M6E; Anti-Nectin 4 ADC ASG-22CE; Anti-nectin-4 Monoclonal Antibody-Drug Conjugate AGS-22M6E; ASG-22CE; Enfortumab Vedotin-ejfv; Padcev
Procedure: MR Urography — Undergo MRU
  Other Names: Magnetic Resonance Urography
Procedure: Nephroureterectomy — Undergo nephroureterectomy
  Other Names: Ureteronephrectomy
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II clinical trial tests how well pembrolizumab plus enfortumab vedotin prior to and after radical nephroureterectomy works in treating patients with high-risk upper tract urothelial cancer. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Enfortumab vedotin (EV) is a monoclonal antibody, enfortumab, linked to an anticancer drug called vedotin. It works by helping the immune system to slow or stop the growth of cancer cells. Enfortumab attaches to a protein called nectin-4 on cancer cells in a targeted way and delivers vedotin to kill them. It is a type of antibody-drug conjugate. Radical nephroureterectomy (RNU) is the surgical removal of a kidney and its ureter. Giving pembrolizumab plus enfortumab vedotin before surgery may make the tumor smaller and may reduce the amount of normal tissue that needs to be removed and giving pembrolizumab after surgery may kill any remaining cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess pathologic objective response rate (ORR; complete response [CR; pT0] and partial response [PR; < pT2] rate) at the time of radical nephroureterectomy.

II. To assess recurrence-free survival post radical nephroureterectomy.

SECONDARY OBJECTIVE:

I. To describe the side effect profile, tolerability, and surgical complications in patients receiving neoadjuvant pembrolizumab (pembro)/ enfortumab vedotin (EV) prior to RNU.

EXPLORATORY OBJECTIVE:

I. Correlative studies will evaluate the predictive potential of imaging and ureteroscopic response (visualization of tumor, biopsy, and cytology), and urinary, serum, and tissue biomarkers to pathologic response.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) and enfortumab vedotin IV on study. Patients undergo radical nephroureterectomy and receive pembrolizumab IV on study Patients also undergo magnetic resonance urogram (MRU) imaging and undergo blood, urine and tissue sample collection throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of high-risk upper tract urothelial carcinoma will be enrolled in this study
* Male participants: A male participant must agree to use a contraception during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period
* Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 6 months after the last dose of study treatment
* Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides. Newly obtained biopsies are preferred to archived tissue
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention
* Absolute neutrophil count (ANC) >= 1500/uL (Specimens must be collected within 10 days prior to the start of study intervention)
* Platelets >= 100000/uL (Specimens must be collected within 10 days prior to the start of study intervention)
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L (Specimens must be collected within 10 days prior to the start of study intervention)
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance [CrCl]) (Specimens must be collected within 10 days prior to the start of study intervention) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN
* Total bilirubin =<1.5 ×ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 × ULN (Specimens must be collected within 10 days prior to the start of study intervention)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase [SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases) (Specimens must be collected within 10 days prior to the start of study intervention)
* International normalized ratio (INR) OR prothrombin time (PT) activated partial thromboplastin time (aPTT) =< 1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (Specimens must be collected within 10 days prior to the start of study intervention)

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

  * Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks [could consider shorter interval for kinase inhibitors or other short half-life drugs] prior to allocation

  * Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible. Participants with endocrine-related AEs grade =< 2 requiring treatment or hormone replacement may be eligible
  * Note: If the participant had major surgery, the participant must have recovered adequately from the procedure and/or any complications from the surgery prior to starting study intervention
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-central nervous system (CNS) disease
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist registered trademark) are live attenuated vaccines and are not allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of Human Immunodeficiency Virus (HIV) infection. However, subjects who are on anti-retroviral therapy, have a viral load < 200 copies/milliliter, and CD4 count > 200/microliter, with a low risk of acquired immunodeficiency syndrome (AIDS)-related outcomes will be considered for enrollment.

  * Note: No HIV testing is required unless mandated by local health authority
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV ribonucleic acid [RNA] is detected) infection. Subjects who have underwent treatment with stable hepatitis B (defined as HBV deoxyribonucleic acid [DNA] < 500 IU/mL) are eligible. Patients with prior curative treatment of Hepatitis C virus are allowed if previously treated > 2 weeks prior to treatment initiation and HCV RNA undetectable by established laboratory values. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has had an allogenic tissue/solid organ transplant
* Subjects who have previously received enfortumab vedotin or other MMAE-based ADCs
* Subjects with an estimated life expectancy < 12 weeks
* Subjects with known severe (>= grade 3) hypersensitivity to any enfortumab vedotin excipient contained in the drug formulation of enfortumab vedotin (including histidine, trehalose dihydrate, and polysorbate 20). Subjects with known severe (>= grade 3) hypersensitivity to any pembrolizumab excipient contained in the drug formulations of pembrolizumab
* Subjects with another underlying medical condition that, in the opinion of the investigator, would impair the ability of the subject to receive or tolerate the planned treatment and follow-up; any known psychiatric or substance abuse disorders that would interfere with cooperating with the requirements of the study
* Subjects with active keratitis or corneal ulcerations. Subjects with superficial punctate keratitis are allowed if the disorder is being adequately treated in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological objective response (ORR) rate | from radical nephroureterectomy through study completion, an average of 1 year
  Will be assessed by the combination of partial response (PR) and complete response (CR). PR is defined as pathologic stage <T2 disease. CR is defined as pT0 disease and assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.
Radiographic recurrence-free survival | From radical nephroureterectomy to 1 year

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post treatment
  Will be assessed using the National Cancer Institute, Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
Rates of completion of neoadjuvant pembrolizumab and enfortumab vedotin | Up to 3 years
  Will be assessed as completion of all infusions of both agents and successful completion of radical nephroureterectomy.
Perioperative complications | Up to 30 days post- radical nephroureterectomy
  Will be assessed based on the Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Chamie, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States